CLINICAL TRIAL: NCT01649518
Title: A Measurement of Knee Osteoarthritis Usual Care
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S54497
Record Dates: First submitted 2012-07-18; First posted 2012-07-25 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2012-06

CONDITIONS: Osteoarthritis, Knee; Guideline Adherence; Quality Indicators, Health Care
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Osteoarthritis is the most common affection of joints worldwide. Multiple international guidelines on the approach and treatment of knee osteoarthritis are available. Nevertheless there seems to be a gap between usual care and the preferred one.

A vigorous set of evidence-based quality indicators on osteoarthritis diagnosis and therapy was developed by a multidisciplinary expert team. This project aims to map usual care and to explore the gaps between usual care and international guidelines in a second stage. This will enable us to develop a tightly targeted quality improvement intervention later on.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee osteoarthritis

Exclusion Criteria:

* Knee replacement surgery
* Acute trauma (recruitment by orthopedic surgeons)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General Practice: Based on the electronic patient files of general practiotioners of the MEDIDOC users-group (an electronic software package) a list will be generated of patients diagnosed with knee osteoarthritis. A random sample of these patients will be addressed to take part into the study by a questionnaire.
  Orthopedic Surgery: Patients, consulting orthopedic surgeons for knee osteoarthritis will receive a patient questionnaire.
  Physiotherapy: Patients, recruited by general practitioners and orthopedic surgeons will be asked about the care they received by their physiotherapist. Moreover physiotherapists will be recruited by the national association of physiotherapists to complete a questionnaire about the care they usually deliver.
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2012-11; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Guideline adherence measured by a number of quality indicators and presented as the percentage of patients in whom a quality indicator was reached | one measurement at the point of recruitment
  Guideline adherence by physicians and physiotherapists will be measured by quality indicators. A questionnaire about the care patients received from diagnosis of knee osteoarthritis till now will be used.

SECONDARY OUTCOMES:
Barriers and facilitators for guideline adherence | 10 years
  Barriers and facilitators for guideline adherence will be explored by focusgroup research with focusgroups of general practitioners, orthopedic surgeons and patients

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium